CLINICAL TRIAL: NCT01126879
Title: Phase 2 Trial of Genistein in Men With Circulating Prostate Cancer Cells
Brief Title: Genistein in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closed due to low accrual
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI 09U2; NCI-2010-00941; STU00019487 (Other: Northwestern University IRB); P50CA090386 (NIH)
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-04

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage II Prostate Cancer; Stage III Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive oral genistein once daily for 3 months beginning at least 1 month prior to radical prostatectomy.
  Interventions: Dietary Supplement: genistein; Procedure: therapeutic conventional surgery
- Arm II (Placebo Comparator): Patients receive an oral placebo once daily for 3 months beginning at least 1 month prior to radical prostatectomy.
  Interventions: Other: placebo; Procedure: therapeutic conventional surgery

INTERVENTIONS:
Dietary Supplement: genistein — Given orally
  Other Names: CI 75610; Genestein; genisteol; genisterin; prunetol; sophoricol
  Arms: Arm I
Other: placebo — Given orally
  Other Names: PLCB
  Arms: Arm II
Procedure: therapeutic conventional surgery — Radical prostatectomy for treatment of prostate cancer

SUMMARY:
RATIONALE: Genistein may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This randomized phase II trial is studying how well genistein works in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether genistein treatment will decrease the number of circulating prostate cells (CPCs) in the peripheral blood as measured by qRT-PCR for PSA performed on RNA extracted from peripheral blood mononuclear cells (PBMNCs).

SECONDARY OBJECTIVES:

I. Determine the natural history of circulating prostate cells (CPCs) in a cohort of subjects prior to and post radical prostatectomy.

II. Compare the measurement of PSA between three separate methods: in CPCs by qRT-PCR, in serum by the standard clinical chemistry assay (i.e., ELISA), and in plasma and serum by the nano-PSA assay.

III. Measure the effect of genistein on gene and protein expression in prostate tissue by qRT-PCR and immunohistochemistry, respectively, for the following genes and their respective protein products: HSP27, MMP-2, ALK-2, BASP1, and HCF2.

OUTLINE:

Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral genistein once daily for 3 months beginning at least 1 month prior to radical prostatectomy.

ARM II: Patients receive oral placebo once daily for 3 months beginning at least 1 month prior to radical prostatectomy.

All patients undergo radical prostatectomy at least 2 weeks, but not more than 3 months following the start of therapy.

After completion of study treatment, patients are followed at 1, 6, and 12 months.

ELIGIBILITY:
Inclusion

* Participants must have a pathologic diagnosis of prostate cancer within the past 6 months, have clinical stage T1-3 disease, PSA >= 10, Gleason score >= 8, and have elected to undergo radical prostatectomy; those found to have detectable circulating prostate cancer cells in the blood as detected by qRT-PCR for PSA will be eligible to proceed onto the treatment phase of the protocol; pathology slides used for diagnosis will be submitted to the SPORE tissue pathology core for review
* ECOG performance status 0-1
* Hemoglobin > 9.0gm/dl
* Platelets >= 100 K/uL
* ANC > 1000/uL
* AST (SGOT)/ALT (SGPT) < 3X upper limit of normal
* Creatinine < 2.0 mg/dl
* Total bilirubin < 2 mg/dl (Note: Subjects with a higher level of bilirubin due to a familial defect in bilirubin metabolism will be considered on an individual basis)
* Participants must agree not to take soy supplements
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to take study agent for at least 2 weeks prior to radical prostatectomy

Exclusion

* History of venous thrombosis within past year
* Participants must not be receiving active therapy for neoplastic disorders (including hormone or radiation therapy for prostate cancer)
* Participants may not be receiving any other investigational agents
* Known soy intolerance
* Medical conditions that, in the opinion of the investigators, would jeopardize either the patient or the integrity of the data obtained

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02-03 (Actual); Primary Completion 2013-05-09 (Actual); Study Completion 2013-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Catalona, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened on October 21, 2010 with an accrual goal of 30 patients with firs the patient enrolled March 3, 2011. The study was designed as a randomized blinded drug/placebo study but was amended to a single arm drug study and accrual reduced to 18. Study closed permanently on May 28, 2014 due to low accrual with 12 patients treated on study.
Pre-assignment Details: Patients entered the study and were treated in a double blinded fashion with a ration of 2:1 Genistein:Placebo. Unblinding occured if it was medically necessary otherwise blinding was maintained until the time of data review.
Groups:
- Arm I - Genistein: Patients receive oral genistein once daily for 3 months beginning at least 1 month prior to radical prostatectomy.
  Genistein: Given orally
  Therapeutic conventional surgery: Radical prostatectomy for treatment of prostate cancer
- Arm II - Placebo: Patients receive an oral placebo once daily for 3 months beginning at least 1 month prior to radical prostatectomy.
  Placebo: Given orally
  Therapeutic conventional surgery: Radical prostatectomy for treatment of prostate cancer
Period: Overall Study
Arm/Group | Arm I - Genistein | Arm II - Placebo
Started | 8 | 4
Started 3 Months of Genistein/Placebo | 8 | 4
Prostatectomy or Radiation | 8 | 4
Completed 3 Months Genistein/Placebo | 4 | 2
Completed | 3 | 2
Not Completed | 5 | 2
Not completed — Progressive Disease | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I - Genistein: Patients receive oral genistein or placebo once daily for 3 months beginning at least 2 weeks prior to radical prostatectomy.
  Genistein: Given orally
  Therapeutic conventional surgery: Radical prostatectomy for treatment of prostate cancer
- Arm II - Placebo: Patients receive oral genistein or placebo once daily for 3 months beginning at least 2 weeks prior to radical prostatectomy.
  Placebo: Given orally
  Therapeutic conventional surgery: Radical prostatectomy for treatment of prostate cancer
- Total: Total of all reporting groups
Arm/Group | Arm I - Genistein | Arm II - Placebo | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 8 | 3 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Circulating Prostate Cells (CPCs) in the Blood as Determined by qRT-PCR for PSA on RNA Extracted From PBMNCs
Description: Blood will be collected to analyze the number of CPC's at screening, after 1-month of treatment, at surgery and at 1 and 12 months after surgery.
Time Frame: At screening, after 1-month of treatment, at surgery and at 1 and 12 months after surgery
Population: Data was not collected for analysis of this endpoint due to the study closing before the accrual goal was met.
Arm/Group | Arm I - Genistein | Arm II - Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Natural History of Circulating Prostate Cells (CPCs) in a Cohort of Subjects Prior to and Post Radical Prostatectomy
Description: Blood will be drawn to analyze the natural history of circulating prostate cells (CPCs) in a cohort of subjects at baseline and 1 and 12 months after surgery.
Time Frame: At baseline, 1 and 12 months after surgery
Population: Data was not collected for analysis of this endpoint due to the study closing before the accrual goal was met.
Arm/Group | Arm I - Genistein | Arm II - Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Measure the Effect of Genistein on Select Gene and Protein Expressions in Prostate Tissue
Description: At baseline and time of surgery, tissue will be collected to measure the effect of genistein on select gene and protein expressions in prostate tissue.
Time Frame: At baseline and at time of surgery
Population: Data was not collected for analysis of this endpoint due to the study closing before the accrual goal was met.
Arm/Group | Arm I - Genistein | Arm II - Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Measurement of PSA in Serum and Plasma by Nanotechnology
Description: Blood will be collected to measure PSA in serum and plasma by nanotechnology at screening, after 1-month of treatment, at surgery and at 1 and 12 months after surgery.
Time Frame: At screening, after 1-month of treatment, at surgery and at 1 and 12 months after surgery
Population: Data was not collected for analysis of this endpoint due to the study closing before the accrual goal was met.
Arm/Group | Arm I - Genistein | Arm II - Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events assessed at the following timepoints for the study: at the start of treatment, at surgery or radiation, at clinic visits occurring 1-3 months post-surgery, or post-initiation of radiation therapy, or at 3 months for those not undergoing surgery or radiation, as well as at a 4 month telephone contact.
Description: Adverse events were collected by patient reports
Arm/Group | Arm I - Genistein | Arm II - Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/4
Other Adverse Events (participants affected / at risk) | 2/8 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I - Genistein (N=8) | Arm II - Placebo (N=4)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I - Genistein (N=8) | Arm II - Placebo (N=4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Large pimple (Skin and subcutaneous tissue disorders) | 0 | 1
Emergency right inguinal repair (Surgical and medical procedures) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0
INR Increased (Investigations) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was closed by an internal safety and data monitoring committee due to slow accrual of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes